CLINICAL TRIAL: NCT00419666
Title: PK and PD of Calcitriol Following Twice Daily Application of Calcitriol 3 µg/g Ointment Under Conditions of Maximal Use in Adolescents With Plaque Psoriasis
Brief Title: A Study of Calcitriol BID Topical Treatment in Adolescents With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.18102
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2019-11

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Calcitriol; Psoriasis; PK; Adolescents
MeSH Terms: conditions — Psoriasis | interventions — Calcitriol

ARMS (1):
- Calcitriol 3mcg/g (Experimental): Participants receive calcitriol 3 micrograms per gram (mcg/g) ointment applied topically twice daily for 56 days.
  Interventions: Drug: Calcitriol 3mcg/g

INTERVENTIONS:
Drug: Calcitriol 3mcg/g — Calcitriol 3mcg/g ointment applied twice daily for 56 weeks.
  Other Names: CD2027; Vectical

SUMMARY:
This is an open-label, multicenter study to assess the systemic exposure to calcitriol in the adolescent population. Calcitriol 3µg/g ointment (2 mg/cm² per application) is to be applied twice daily to involved skin (10 - 35% BSA involved, excluding face, scalp and intertriginous areas) for 56 days (8 weeks). Full Pharmacokinetic (PK) and Pharmacodynamic (PD) profile will be collected during the first 3 weeks of the study; safety and efficacy data will be collected for the 8 weeks of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis
* 10 - 35% BSA of involved skin
* Age 12 - 17

Exclusion Criteria:

* Other type of psoriasis (other than plaque)
* Significant abnormal lab findings
* Vit D insufficiency

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2009-09-24 (Actual); Study Completion 2009-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (7):
- United States (5):
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Children's Hospital, Department of Pediatric and Adolescent Dermatology, San Diego, California
  - Dermatology Center For Children & Young Adults, Eagan, Minnesota
  - University of Texas-Houston Medical Center Dept of Dermatology, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
- Canada (2):
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Newlab Clinical Research, Inc., St. John's, Newfoundland and Labrador

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 7 sites (5 in United States and 2 in Canada) between 01 Aug 2006 (first participant enrolled) to 24 Sep 2009 (last participant completed).
Pre-assignment Details: A total of 25 participants were enrolled and completed the study.
Groups:
- Calcitriol 3mcg/g: Participants received calcitriol 3 micrograms per gram (mcg/g) ointment applied topically twice daily for 56 days.
Period: Overall Study
Arm/Group | Calcitriol 3mcg/g
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population consisted of all participants who were enrolled and to whom medication was dispensed.
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.7 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 16
  Race: Black | 2
  Race: Asian | 1
  Race: Hispanic | 4
  Race: Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Trough Plasma Levels (Ctrough) of Calcitriol
Description: Trough plasma levels (Ctrough) of calcitriol was reported.
Time Frame: Day 0 (Baseline), Day 14, Day 21, and Day 56
Population: Safety population consisted of all participants in the ITT population who had applied the study medication at least once.
Measure: Mean (Standard Deviation); unit: Picograms Per Millilitre (pg/mL)
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
Picograms Per Millilitre (pg/mL)
  Day 0 (Baseline) | 65.04 (18.851)
  Day 14 | 62.53 (17.742)
  Day 21 | 61.87 (17.703)
  Day 56 | 61.46 (22.811)

2. Primary Outcome: The Observed Peak Drug Concentration (Cmax) of Calcitriol
Description: Cmax of calcitriol was reported.
Time Frame: Day 0 (Baseline), Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
pg/mL
  Day 0 (Baseline) | 75.74 (24.337)
  Day 21 | 73.18 (21.514)

3. Primary Outcome: Area Under the Concentration-Time Curve From Pre-Application (T0) Through 9 Hours Post Dosing (AUC [0-9 Hours])
Description: The AUC(0-9 hours) that is area under the plasma concentration-time curve from time 0 to 9 hours after dosing was reported.
Time Frame: 0 (predose) and 9 hours post dose on Day 0 (Baseline), Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picograms. hours per millilitre(pg.h/mL)
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
Picograms. hours per millilitre(pg.h/mL)
  Day 0 (Baseline) | 575.12 (181.761)
  Day 21 | 549.29 (155.277)

4. Primary Outcome: Area Under the Concentration-Time Curve From Pre-Application (T0) Through 12 Hours Post Dosing (AUC [0-12 Hours])
Description: The AUC(0-12 hours) that is area under the plasma concentration-time curve from time 0 to 12 hours after dosing was reported.
Time Frame: 0 (predose) and 12 hours post dose on Day 0 (Baseline), Day 21
Population: Safety population consisted all participants in the ITT population who had applied the study medication at least once.
Measure: Mean (Standard Deviation); unit: pg.h/mL
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
pg.h/mL
  Day 0 (Baseline) | 764.74 (230.003)
  Day 21 | 737.74 (203.740)

5. Primary Outcome: Time at Which Maximum Concentration (Cmax) Occurred (Tmax)
Description: Tmax is the time to reach maximum concentration and was reported for calcitriol.
Time Frame: Day 0 (Baseline), Day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
hours
  Day 0 (Baseline) | 4.00 [0.0 to 9.0]
  Day 21 | 3.97 [0.0 to 9.0]

6. Secondary Outcome: Change From Baseline in Effect of Calcitriol Ointment on Calcium (Serum Calcium, Urinary (U) Calcium Random) and Phosphorus Homeostasis up to Day 56
Description: Calcium homeostasis was analyzed with serum calcium albumin adjusted, serum calcium, urinary calcium/creatinine ratio, urinary (U) calcium random as parameters. Phosphorus homeostasis was analyzed with phosphorus as parameter. Change from baseline in the effect of calcitriol ointment on calcium (serum calcium, U calcium random) and phosphorus homeostasis up to Day 56 was reported.
Time Frame: From baseline (Day 0) up to Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (Mg/dL)
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
milligrams per deciliter (Mg/dL)
  Serum Calcium | 0.08 (0.254)
  Urinary (U) Calcium Random | 1.00 (6.767)
  Phosphorus | 0.20 (0.641)

7. Secondary Outcome: Change From Baseline in Effect of Calcitriol Ointment on Calcium (Serum Calcium Albumin Adjusted) Homeostasis up to Day 56
Description: Calcium homeostasis was analyzed with serum calcium albumin adjusted, serum calcium, urinary calcium/creatinine ratio, urinary (U) calcium random as parameters. Change from baseline in the effect of calcitriol ointment on calcium (serum calcium albumin adjusted) homeostasis up to Day 56 was reported.
Time Frame: From baseline (Day 0) up to Day 56
Population: Safety population consisted all participants in the ITT population who had applied the study medication at least once.
Measure: Mean (Standard Deviation); unit: Millimoles Per Litre (mmol/L)
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
Millimoles Per Litre (mmol/L) | -0.01 (0.083)

8. Secondary Outcome: Change From Baseline in Effect of Calcitriol Ointment on Calcium (Urinary Calcium/Creatinine Ratio) Homeostasis up to Day 56
Description: Calcium homeostasis was analyzed with serum calcium albumin adjusted, serum calcium, urinary calcium/creatinine ratio, urinary (U) calcium random as parameters. Change from baseline in the effect of calcitriol ointment on calcium (urinary calcium/creatinine ratio) homeostasis up to Day 56 was reported.
Time Frame: From baseline (Day 0) up to Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
Ratio | 0.01 (0.076)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was any unfavorable and unintended sign (including an abnormal laboratory finding assessed as clinically significant and different from the baseline visit), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Number of participants with adverse events were reported.
Time Frame: From start of the study to Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calcitriol 3mcg/g
Number analyzed (Participants) | 25
Participants | 13

ADVERSE EVENTS:
Time Frame: From start of the study to Day 56
Arm/Group | Calcitriol 3mcg/g
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcitriol 3mcg/g (N=25)
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other